CLINICAL TRIAL: NCT02891733
Title: Retrospective Analysis of the Expression of the Neurotensin Receptor by Metastatic Lung Adenocarcinomas
Acronym: NTS
Status: Withdrawn | Type: Observational
Why Stopped: The principal investigator decided to stop the study.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: NTS
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Lung Adenocarcinomas
Keywords: Expression of the Neurotensin; Neurotensin
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is the leading cause of cancer mortality in France and worldwide. 60% of patients present themselves with a disease diagnosis immediately metastatic non curable. Adenocarcinomas account for 50% of incident tumors. Treatment is based on the platinum-based chemotherapy with or without maintenance therapy. When there is to exhaust this first line, a second line treatment is offered to the patient. Three drugs are allowed in this situation: docetaxel, erlotinib (inhibitor of the tyrosine kinase activity of the receptor for epidermal growth factor - TKI-EGFR) and pemetrexed (which in fact has become virtually standard in first online and in combination with platinum in all patients with non-squamous cancer, so that his place is in second line reduced facto). There is no recommendation for treatment in third line situation where only erlotinib is allowed.

Most recently, the nivolumab, anti-PD1 monoclonal antibody (which aims to enable immunutaire system) saw its demonstrated effectiveness in the second line and beyond in the two Phase 3 trials where it was compared with docetaxel for the treatment of squamous cell carcinoma and non-squamous. The very recent availability in France of the drug under an ATU fact that it will most likely become a standard second line, which will tend to place the third line docetaxel.

Therefore, erlotinib will be in 4th line situation. However, in the absence of an EGFR mutation (which is only seen in more than 10% of Caucasian patients) use of the drug does not seem appropriate or even harmful. A selection of patients likely to benefit from the prescription of EGFR TKI-is essential.

Neurotensin (NTS) is a polypeptide of 13 amino acids present and active in the central nervous system and the periphery. At the peripheral level, neurotensin is secreted postprandial by endocrine cells in the intestinal mucosa and is involved in the motor functions of the gastrointestinal tract. The effects of neurotensin pass through the activation of three subtypes of receptors which, mainly, NTSR1 and NTSR2 which are receptors coupled to G proteins in the extra-digestive normal tissues, including lung, torque NTS / NTSR1 n is not expressed physiologically. Rather, this complex is likely to recur in tumor tissues.

The mechanism of this effect is derogatory activation torque NTS / NTSR1 of matrix metalloproteinases which causes the release by the cell membrane ligands "EGF-like" and thus, activation of HER receptor (EGFR or HER1, HER2 and HER3). Indeed, in experimental tumors created by subcutaneous injection in athymic mouse cell lines adenocarcinomas NTS + / NTSR1 + (non-mutated EGFR), treatment with erlotinib - which blocks EGFR pathway - causes a significant decrease of tumor growth.

Expression of the neurotensin receptor in cancer cells metastatic primary bronchial adenocarcinoma is not known. Therefore, its pejorative prognostic value is not confirmed in the metastatic setting.

DETAILED DESCRIPTION:
The objectives of this work purely descriptive, are:

* Evaluate the expression by tumor cells of the neurotensin receptor on a retrospective series of patients:
* Consecutively treated between 2010 and 2015 at St. Joseph hospital (about a hundred patients) and the Saint-Antoine hospital (three hundred patients), holders of a metastatic and primary lung adenocarcinoma having received all even first-line chemotherapy with a platinum agent (cisplatin or carboplatin) and pemetrexed (Alimta °)
* If possible, the records of patients treated at St. Joseph Hospital and Saint-Antoine Hospital between 2005 and 2010 as part of clinical trials evaluating the value of erlotinib will also be sought,
* Develop a score expression NTSR1 taking into account the percentage of tumor cells expressing the receptor and the intensity of the marking,
* Correlate labeling cells by NTSR1 with the clinical course of patients to see if expression NTSR1 is a factor of poor prognosis in metastatic patients.

Teams involved:

Services:

* Pharmacy that will establish the list of patients have been treated with the same chemotherapy,
* Pathological anatomy-to group blades and ensure immunohistochemical staining and reading,
* Pneumology and Thoracic Oncology to resume the clinical history of patients.

The scientific coordination of the study will be conducted by INSERM UMR-S 1007, cellular homeostasis and cancer - Reprogramming of biological and alternative therapies responses (University Center of the Holy Fathers, 45 rue des Saints Pères, 75006 Paris), one team under the direction of Dr. Patricia Forge, working on the couple NTS / NTSR1.

expected benefits

Beyond two or three conventional chemotherapy line, which will no doubt add - for a proportion of patients still to be determined - the new immunotherapy drugs, there is no longer any recommendations for treatment of patients lung cancer metastatic non-small cells. Erlotinib is an option since there is no limitation in its approval of prescription ond line. However, in the absence of EGFR mutation, the therapeutic value of the drug appears to be very low. Preclinical data that investigators obtained in the laboratory are hypothesize that tumors expressing NTSR1 could meet the same TKI EGFR in the absence of mutation in the receptor. The planned study will assess the percentage of patients in this situation in order to prepare the organization of a Phase II study to evaluate the clinical relevance of a TKI EGFR in this selected population of patients carrying of a non-mutated tumor.

Nature of the data collected

A file will be drawn from the clinical data found in files: all patients are carriers of metastatic primary lung adenocarcinoma and having all received the same chemotherapy.

The data obtained will be: age, sex, smoking status, number of courses of chemotherapy received and the response to treatment, the usual chronological parameters for the establishment of the survival curves. Histological samples will be processed locally in each of the two hospitals, according to a specific procedure to be determined between laboratories and INSERM Unit.

Identification of subjects and circulation and processing of data

In this study, the inclusions are carried out within the hospital group Paris Saint-Joseph and Saint-Antoine hospital. Histological samples will be processed locally in each of the two hospitals, according to a specific procedure to be determined between pathological anatomy and INSERM Unit Laboratories.

These histological samples will be stored at the Pathological Anatomy Laboratory Groupe Hospitalier Paris Sani Joseph.

Each study participant will be identified by a code of inclusion (first name and surname - year of birth). The concordance table to link the assigned code and the participant's name will be kept in each of the participating centers, in a file protected by a password specific to the principal investigator of each center. Data collected from different centers on anonymous paper media (only the code for inclusion of each patient are included) will be centralized within the GHPSJ and entered in a database which anonymous access is protected by the PIN each in the study of GHPSJ. Data processing and statistical analysis will be performed on the GHPSJ site in collaboration with the Clinical Research Unit of the European Hospital Georges Pompidou.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma in metastatic stage
* Patients received
* The same first-line chemotherapy with a platinum agent (cisplatin or carboplatin) and pemetrexed (Alimta °)

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consecutively treated between 2010 and 2015 at St. Joseph hospital (about a hundred patients) and the Saint-Antoine hospital (three hundred patients), holders of a primary lung adenocarcinoma in the metastatic setting and having all received the same first-line chemotherapy with a platinum agent (cisplatin or carboplatin) and pemetrexed (Alimta °)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patient expressing Neurotensin receptor ( NTSR1) in their tumor | Day 1

IPD SHARING:
Plan to Share IPD: Undecided